CLINICAL TRIAL: NCT04453397
Title: A Single Patient Protocol for TNB-383B, a Bispecific Antibody Targeting BCMA in a Subject With Relapsed/Refractory Multiple Myeloma
Brief Title: Expanded Access for TNB-383B in a Subject With Relapsed/Refractory Multiple Myeloma
Status: No longer available | Type: Expanded Access
Sponsor: TeneoOne Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TNB383B.9001
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: TNB-383B — TNB-383B is a bispecific antibody targeting BCMA on tumor cells and CD3 on T-cells.

SUMMARY:
This is a single patient protocol for TNB-383B in a subject with relapsed/refractory multiple myeloma (MM) who is not a candidate for treatment regimens known to provide clinical benefit in MM.

ELIGIBILITY:
Inclusion Criteria:

* Adequate bone marrow function
* eGFR ≥ 30 mL/min
* Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
* Serum calcium (corrected for albumin) at or below the ULN range

Exclusion Criteria:

* Candidate for treatment regimens known to provide clinical benefit in MM
* Active infection requiring parenteral anti-infective treatment
* Any medical or psychiatric condition which in the opinion of the investigator or Teneobio Medical Monitor places the subject at an unacceptably high risk for toxicities, could interfere with successful or safe delivery of therapy, or could interfere with evaluation of the investigational product or interpretation of subject safety

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ben Buelow, Study Chair — Amgen
Locations (1):
- Wake Forest, Winston-Salem, North Carolina, United States